CLINICAL TRIAL: NCT05061485
Title: The Effect of Macronutrients on Fibroblast Growth Factor 21 (FGF21) Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: The FGF21-macro study
Record Dates: First submitted 2021-09-09; First posted 2021-09-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — Sucrose; Proteins; CD36 Antigens

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sucrose (Experimental): The participants will be served a test drink with 75g sucrose dissolved in water
  Interventions: Other: Sucrose
- Sucrose + protein (Experimental): The participants will be served a test drink with 75g sucrose dissolved in water and ~ 100 kcal protein (whey protein)
  Interventions: Other: Sucrose + protein
- Sucrose + fat (Experimental): The participants will be served a test drink with 75g sucrose dissolved in water and ~ 100 kcal fat (cream)
  Interventions: Other: Sucrose + fat

INTERVENTIONS:
Other: Sucrose — The participants consume A) water with 75 g sucrose
  Arms: Sucrose
Other: Sucrose + protein — The participants consume B) water with 75 g sucrose + approx. 100 kcal protein
  Arms: Sucrose + protein
Other: Sucrose + fat — The participants C) water with 75 g sucrose + approx. 100 kcal fat
  Arms: Sucrose + fat

SUMMARY:
The aim of this randomized cross-over study is to investigate how consumption of protein and fat affects the FGF21 response triggered by sucrose. The hypothesis is that the consumption of protein, but not fat, will attenuate the FGF21 response triggered by sucrose.

Exploratory, and in order to investigate mechanisms behind the potential attenuation in the sucrose-induced FGF21 response after protein consumption, glucose, insulin, glucagon, triglycerides, amino acids, glicentin and cholecystokinin (CCK) will be assessed before and after consumption of sucrose, sucrose+protein and sucrose+fat. Furthermore, the association between the FGF21 response after consumption of sucrose, sucrose + protein and sucrose + fat and subjective rating of appetite for sweet will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Caucasian
* Healthy men and women
* Age between 18-50 years
* Body mass index (BMI) between 20-27 kg/m2

Exclusion Criteria:

* Chronic diseases or significant health problems that are disruptive for participation in the study (as judged by the principal investigator/clinical responsible)
* Use, currently or within the previous 3 months, of medication that has the potential of affecting any of the blood parameters assessed in the study (as judged by the principal investigator/clinical responsible)
* Blood donation within the last 3 months or during the study period
* Smoking, smoking cessation within the past 3 months, or nicotine use (electronic cigarettes, gum, etc.)
* Currently dieting or having lost/gained a significant amount of weight (±3 kg) in the previous 3 months
* Women who are pregnant, breast-feeding or have the intention of becoming pregnant during the study period
* Food allergies or food intolerance relevant for the study
* Substance abuse (within the last 12 months)
* Alcohol intake above the recommendations from the Danish Health and Medicines Authority
* Simultaneous participation in other clinical studies that can interfere with the current study
* Inability, physically or mentally, to comply with the procedures required by the study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Difference in FGF21 concentration after consumption of sucrose vs. sucrose+protein | Difference in plasma concentration of FGF21 between two test days
  Difference (pg/ml) in plasma FGF21 concentration after consumption of sucrose vs. sucrose+protein. Concentration of FGF21 is measured at time 0 and 60, 120, 180, and 240 min after consuming the test drinks.

SECONDARY OUTCOMES:
Difference in FGF21 concentration after consumption of sucrose vs. sucrose+fat | Difference in plasma concentration of FGF21 between two test days
  Difference (pg/ml) in plasma FGF21 concentration after consumption of sucrose vs. sucrose+fat. FGF21 is measured at time 0 and 60, 120, 180, and 240 min after consuming the test drinks.
Difference in glucose concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. | Difference in plasma concentration of glucose between the three test days
  Difference (mmol/l) in plasma glucose concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. Glucose is measured at time 0 and 60, 120, 180, and 240 min after consuming the test drinks.
Difference in insulin concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. | Difference in serum concentration of insulin between the three test days
  Difference (pmol/l) in serum insulin concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. Insulin is measured at time 0 and 60, 120, 180, and 240 min after consuming the test drinks.
Difference in glucagon concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. | Difference in plasma concentration of glucagon between the three test days
  Difference (pg/ml) in plasma glucagon concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. Glucagon is measured at time 0 and 60, 120, 180, and 240 min after consuming the test drinks.
Difference in triglyceride concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. | Difference in serum concentration of triglycerides between the three test days
  Difference (mmol/l) in serum triglyceride concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. Triglyceride is measured at time 0 and 60, 120, 180, and 240 min after consuming the test drinks.
Difference in amino acid concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. | Difference in serum concentration of amino acids between the three test days
  Difference in serum amino acid concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. Amino acids are measured at time 0 and 60, 120, 180, and 240 min after consuming the test drinks.
Difference in glicentin concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. | Difference in plasma glicentin between the three test days
  Difference (pmol/l) in plasma glicentin concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. Glicentin is measured at time 0 and 60, 120, 180, and 240 min after consuming the test drinks.
Difference in CCK concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. | Difference in plasma CCK between the three test days
  Difference (pmol/l) in plasma CCK concentration after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. CCK is measured at time 0 and 60, 120, 180, and 240 min after consuming the test drinks.
Difference in appetite for sweet after consumption of sucrose vs. sucrose+protein vs. sucrose+fat. | Difference in appetite for sweet between the three test days
  Difference in appetite for sweet is measured using visual analog scales (VAS). The VAS consists of a 100 mm horizontal unbroken line with words anchored at each end describing the extremes. The participants respond to the question asked by placing a vertical mark through the horizontal line corresponding to their perceived feeling at that particular time. Appetite for sweet is assessed at time 0 and 30, 60, 120, 180, and 240 min after consuming the test drinks.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Gillum, Principal Investigator — Novo Nordisk Foundation Center for Basic Metabolic Research, Health and Medical Sciences, University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ramne S, Duizer L, Nielsen MS, Jorgensen NR, Svenningsen JS, Grarup N, Sjodin A, Raben A, Gillum MP. Meal sugar-protein balance determines postprandial FGF21 response in humans. Am J Physiol Endocrinol Metab. 2023 Nov 1;325(5):E491-E499. doi: 10.1152/ajpendo.00241.2023. Epub 2023 Sep 20. PMID 37729024